CLINICAL TRIAL: NCT06051721
Title: A Phase 2a, Randomized, Double-Blind, Active-Controlled Study to Assess the Preliminary Clinical Efficacy, Safety, Tolerability, and Pharmacokinetics, of CYB004 in Participants With Generalized Anxiety Disorder (GAD)
Brief Title: A Study of a N, N-dimethyltryptamine (DMT) Analog (CYB004) in Participants With Generalized Anxiety Disorder (GAD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cybin IRL Limited (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYB004-002
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; GAD; Depression; CYB004; CYB004-002; Psychedelic; DMT; N, N-dimethyltryptamine
MeSH Terms: conditions — Generalized Anxiety Disorder; Depression | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Active (Experimental): Arm A participants will receive a full dose of CYB004 in 2 of 2 medicine sessions, approximately three weeks apart. All participants will receive supportive EMBARK psychotherapy throughout the study.
  Interventions: Drug: CYB004; Behavioral: Psychotherapy
- Arm B: Control (Active Comparator): Arm B participants will receive a low dose of CYB004 in 2 of 2 medicine sessions, approximately three weeks apart. All participants will receive supportive EMBARK psychotherapy throughout the study.
  Interventions: Drug: CYB004; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: CYB004 — CYB004 is a synthetic deuterated N, N-Dimethyltryptamine (DMT) analog.
Behavioral: Psychotherapy — Manualized psychotherapy (called EMBARK) performed by facilitators

SUMMARY:
The purpose of this proof-of-concept trial is to examine the safety, tolerability, and pharmacokinetics (PK), and preliminary clinical efficacy of CYB004 participants with GAD.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 65 years, inclusive, at Screening.
* Has a diagnosis of GAD (as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition [DSM-V] of moderate to severe degree), established through a full psychiatric work up.
* Has a BMI of 18 to 40.0 kg/m2, inclusive at Screening.
* Has been on a stable dose of antidepressant/anxiolytic medication (no more than 50% change) in the last month prior to Screening and has had an inadequate response, as judged by the Investigator.
* Is willing to refrain from taking any benzodiazepines for 5 days or buspirone (or other 5-HT1A agonist) during the 24 hours preceding each dosing visit.
* Provision of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Has a primary DSM-5 psychiatric diagnosis other than GAD within the past 6 months established through a full psychiatric work-up. A secondary diagnosis of MDD may be permissible.
* Current or previously diagnosed schizophrenia spectrum or other psychotic disorders, including schizophrenia, schizoaffective disorder, schizotypal disorder, schizophreniform disorder, brief psychotic disorder or borderline personality disorder; current or previous history of psychosis or bipolar disorder.
* Currently taking a monoamine oxidase inhibitor, tricyclic antidepressant, trazadone, mirtazapine, or a mood stabilizer (including lithium) or has taken any of these medications in the last 3 weeks of trial participation.
* Currently taking antipsychotic medication which are 5-HT2 antagonists or has taken such medication in the last 3 weeks of trial participation.
* Clinically significant risk of suicidality, as determined through a comprehensive psychiatric interview.
* Clinically relevant history of abnormal physical health interfering with the study as determined by medical history and physical examinations obtained during Screening as judged by the Investigator (including [but not limited to], neurological, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder).
* Currently receiving treatment for hypertension or arrhythmia.
* Clinically relevant abnormal laboratory results.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Any other concomitant disease or condition that could interfere with, or for which the treatment might interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this trial.
* Has a presence or relevant history of any organic brain disorders (e.g., epilepsy, seizure, intracranial hypertension, intracranial bleed and aneurysmal disease, brain tumor or other medical conditions associated with seizures or convulsions).
* Consumes excessive amounts of caffeine (e.g., coffee, tea, caffeinated sodas) or (methyl) xanthines (e.g., chocolate) based on the Investigator's determination and discretion.
* Positive urine test for drugs of abuse or alcohol breath test at Screening or Day 1. A positive test for cannabinoids (e.g. marijuana) at Screening may not exclude a participant if after discussion with and evaluation by the Investigator, the participant agrees not to use any marijuana or other cannabinoid products during the study, and if allowed to participate, the participant must test negative for cannabinoids on Day 1 and Day 22.
* Has participated in a clinical trial and has received a medication or a new chemical entity within 3 months prior to dosing of current study medication.
* Known sensitivity to DMT or ayahuasca.
* Is taking a prescription medicine (except for stable chronic dose of antidepressant/anxiolytic medication(s), sedatives/hypnotics, and hormonal contraceptives or hormonal replacement medications, if applicable), certain herbal supplements (to be reviewed by the Investigator), or over-the-counter (OTC) medicine during the 28 days before dosing.
* Is taking or has taken over the counter (OTC) doses of 5-hydroxytryptophan or St John's Wort within 28 days prior to receiving the study drug.
* Donation of blood or plasma of >400 mL within 1 month prior to first dosing until 4 weeks after final dosing.
* For participants capable of producing sperm: Is not willing to abstain from sperm donation between first dosing and 3 months after final dosing.
* For participants capable: Is pregnant, breastfeeding or planning to conceive.
* Not fluent in the English language.
* Other eligibility considerations (i.e., participant personal circumstances, behavior, and/or any current problem that might interfere with participation or that is incompatible with establishment of rapport or safe exposure to the study drug), as judged by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | Screening (Day-63 and Day-1), Day 2, Day 8, Day 21, Day 23, Day 29, Day 43, Day 64, Day 85, Day 169, Day 266, and End of Treatment (Day 364)
  The HAM-A is a 14-item scale that is used to rate the severity of symptoms of anxiety. Each of the 14 items is defined by a series of symptoms and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Items are scored from 0 (not present) to 4 (very severe), for a total score ranging from 0 to 56. Scores <17 indicate mild anxiety, scores of 18 to 24 indicate mild to moderate anxiety, and scores of 25 to 30 or higher indicate moderate to severe anxiety.

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | Screening (Day-63 and Day-1), Day 2, Day 8, Day 21, Day 23, Day 29, Day 43, Day 64, Day 85, Day 169, Day 266, and End of Treatment (Day 364)
  The HAM-D is a validated 17-item questionnaire administered by the clinician used to assess severity of, and change in, depressive symptoms in the past week. The questionnaire assesses core symptoms of depression, anxiety, and side effects of drug treatment on a scale of 0 to 50 with higher scores indicating more severe depression. Scores of 0-7 are considered normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression (Zimmerman et al., 2013); the maximum score being 52 on the 17-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Inamdar, MBBS, DNB, MFPM, Study Director — Cybin IRL Limited
Locations (6):
- United States (6):
  - Research Centers of America, Hollywood, Florida
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - CenExel ACMR, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Cedar Clinical Research, Murray, Utah

IPD SHARING:
Plan to Share IPD: No